CLINICAL TRIAL: NCT02423083
Title: Phase I Study of Oral Guanabenz for Multiple Sclerosis
Brief Title: Oral Guanabenz for Multiple Sclerosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150117; 15-N-0117
Record Dates: First submitted 2015-04-21; First posted 2015-04-22 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2017-10-30

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis
Keywords: Neuroprotection; Multiple Sclerosis; Clinical Trial; Safety and Tolerability
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Guanabenz

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Drug: Guanabenz

INTERVENTIONS:
Drug: Guanabenz

SUMMARY:
Background:

- People with multiple sclerosis (MS) get lesions in their brain and spinal cord. These cause neurological symptoms and sometimes disability. Researchers want to see if a blood pressure drug called guanabenz can repair lesions and help people with MS.

Objective:

- To see if guanabenz is safe and well tolerated in people with MS.

Eligibility:

- People 18 55 years old with MS who have taken glatiramer acetate for the past year.

Design:

* Participants will be screened in a separate protocol. For 2 months, they will be examined and have magnetic resonance imaging (MRI) scans. This will decide if they are in the Stable or Active MS study group.
* The study will last 5 months. There will be up to 11 visits, 5 overnight.
* Visit 1: overnight stay at the clinic:
* Medical history and physical exam.
* Health questionnaire
* Bladder ultrasound scan
* Brain MRI
* Electrocardiogram (EKG) to measure heart electrical activity
* Blood will be drawn through an intravenous (IV) line.
* Participants may have tests of strength, muscle tone, and movement.
* They will get their first dose of the study drug, a tablet taken once a day.
* Participants will take the study drug at home and keep a medicine diary.
* The dose will slowly increase. Each time, participants will stay overnight at the clinic. They will have a physical exam, EKG, MRI, and IV blood draw.
* Visit 6: Participants will have a physical exam, MRI, and blood drawn. They will get a schedule to slowly lower their drug dose and stop taking guanabenz.
* Participants will have 2 final visits. They will have a physical exam, EKG, MRI, and IV blood draw.

DETAILED DESCRIPTION:
OBJECTIVE:

This Phase 1 clinical study will aim to determine whether therapeutically adequate dosages of guanabenz are safe and well tolerated in patients with multiple sclerosis (MS). It will further provide pharmacokinetic data important for determination of optimal dosing schedule for possible future Phase 2 study.

STUDY POPULATION:

Six patients, ages between 18-55 inclusive, and diagnosis of definite multiple sclerosis by 2010 Revised McDonald Diagnostic Criteria (Polman et al, 2010) will be enrolled. All patients will have been on treatment with glatiramer acetate, a Food and Drug Administration (FDA) approved disease-modifying therapy, for a minimum of year. Four of the patients will be clinically stable with no clinical relapse in the preceding year and no evidence of active inflammation by MRI during the 2-month screening period; 2 patients will be selected based on evidence of on-going, active inflammation seen by MRI during the screening period.

DESIGN:

In this open-label, single site, dose escalation study, the maximum tolerated dose (MTD) of guanabenz in MS patients will be determined. Patients will be screened for participation under the existing MS natural history study 89-N-0045. Sequential patient enrollment will be spaced at least 6 weeks apart. Five study drug doses will be explored: 4mg, 8mg, 16mg, 32mg and 64mg. Dose escalation will ensue if the preceding dose is tolerated, defined both by patient-reported outcomes and objective clinical and imaging assessments. Patients will be maintained on lower doses (4mg-16mg) for 14 days and on higher doses (32 and 64mg) for 28 days.

OUTCOMES:

The primary outcome is MTD, defined as the maximum dose that produces dose-limiting toxicity (DLT) in at most 2 out of the 6 participants. Secondary outcomes include patient-reported outcomes, objective clinical and imaging assessments at 32mg and 64mg, and pharmacokinetics.

ELIGIBILITY:
* INCLUSION CRITERIA:
* MS as defined by the 2010 Revised McDonald MS Diagnostic Criteria (19)
* Age 18-55, inclusive, at the time of the first screening baseline visit
* EDSS 1.0 to 6, inclusive, at the time of the first screening baseline visit
* Able to provide informed consent
* Willing and able to participate in all aspects of trial design and follow-up
* Undergoing treatment with glatiramer acetate for a period of at least 1 year prior to enrollment in the study
* For female patients, agreeing to commit to the use of a reliable/accepted method of birth control (i.e. hormonal contraception, including

birth control pills, injected hormones, and vaginal ring; intrauterine device; barrier methods with spermicide, including diaphragm and condom; or surgical sterilization, including hysterectomy, tubal ligation, and vasectomy) for the duration of the study

ADDITIONAL INCLUSION CRITERION FOR ACTIVE MS COHORT

-Development of new T2 hyperintense or contrast enhancing lesions by MRI during the screening phase, but 3 such lesions on any single scan

EXCLUSION CRITERIA:

* Alternative diagnoses that better explain neurological disability and MRI findings
* Clinically significant medical condition that, in the best judgment of the investigators, may expose the patient to undue risk of harm or prevent the patient from completing the study (examples include, but are not limited to, cerebrovascular disease, substance abuse, ischemic cardiomyopathy, clotting disorder, brittle diabetes, neurodegenerative disorder)
* Undergoing treatment with medications that may interact with guanabenz, including anti-hypertensive agents and/or agents leading to increase in catecholamines (such as tricyclic antidepressants and monoamine oxidase inhibitors)
* Medical contraindication to MRI
* Determination, in the best judgment of the investigators, of the need to treat a prospective participant with steroids for management of MS during the screening period
* Pregnant or breastfeeding woman
* Abnormal screening/baseline blood tests exceeding any of the limits defined below:

A) Serum alanine transaminase or aspartate transaminase levels greater than 3 times the upper limit of normal values

B) Total white blood cell count < 3000/mm3

C) Platelet count < 85000/mm3

D) Serum creatinine level > 2.0 mg/dl and eGFR (estimated glomerular filtration rate) < 60

ADDITIONAL EXCLUSION CRITERIA FOR STABLE MS COHORT

* Evidence of 1 or more clearly documented MS relapses within the last 1 year
* Development of more than 2 lesions per year relative to an MRI performed at least one year before the first screening MRI (the prior MRI can be an outside MRI)
* Development of new T2 hyperintense or contrast-enhancing lesions by MRI during the screening phase

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2015-04-21; Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 3.5 months

SECONDARY OUTCOMES:
Pharmacokinetics of guanabenz in MS patients | 3.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Irene CM Cortese, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lin W, Popko B. Endoplasmic reticulum stress in disorders of myelinating cells. Nat Neurosci. 2009 Apr;12(4):379-85. doi: 10.1038/nn.2273. Epub 2009 Mar 15. PMID 19287390
- [Background] Lin W, Kunkler PE, Harding HP, Ron D, Kraig RP, Popko B. Enhanced integrated stress response promotes myelinating oligodendrocyte survival in response to interferon-gamma. Am J Pathol. 2008 Nov;173(5):1508-17. doi: 10.2353/ajpath.2008.080449. Epub 2008 Sep 25. PMID 18818381
- [Background] Lin W, Lin Y, Li J, Fenstermaker AG, Way SW, Clayton B, Jamison S, Harding HP, Ron D, Popko B. Oligodendrocyte-specific activation of PERK signaling protects mice against experimental autoimmune encephalomyelitis. J Neurosci. 2013 Apr 3;33(14):5980-91. doi: 10.1523/JNEUROSCI.1636-12.2013. PMID 23554479
- [Derived] Clayton BLL, Popko B. Endoplasmic reticulum stress and the unfolded protein response in disorders of myelinating glia. Brain Res. 2016 Oct 1;1648(Pt B):594-602. doi: 10.1016/j.brainres.2016.03.046. Epub 2016 Apr 4. PMID 27055915